CLINICAL TRIAL: NCT01908348
Title: Pilot Study: Dose Dependent Effects of Erythritol on Endothelial Function in Patients With Type 2 Diabetes Mellitus
Brief Title: Dose-Dependent Effects of Erythritol on Endothelial Function in Type 2 Diabetes Mellitus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston University (Other)
Collaborators: Cargill (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: H-32353
Record Dates: First submitted 2013-07-23; First posted 2013-07-25 (Estimated); Last update posted 2018-02-28 (Actual); Status verified 2018-02

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Erythritol; Endothelial function
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Erythritol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Erythritol (Experimental): Orange-flavored beverage containing 6, 12, or 18 grams of erythritol
  Interventions: Dietary Supplement: Erythritol

INTERVENTIONS:
Dietary Supplement: Erythritol

SUMMARY:
This study is an open-label pilot designed to examine the dose-dependent effects of erythritol, a zero calorie sweetener, on endothelial function. Twenty-four subjects with type 2 diabetes mellitus will make three study visits. At each visit, the will consume an orange-flavored beverage containing escalating amounts of erythritol (6, 12, and 18 grams). Endothelial function will be assessed before and two hours after beverage consumption. Endothelial function will be measured as the change in pulse amplitude in response to reactive hyperemia measured in the fingertip by peripheral arterial tonometry. The results will be used to plan a randomized, placebo-controlled study.

ELIGIBILITY:
Inclusion Criteria:

* Male and Female subjects
* Otherwise healthy patients with Type 2 diabetes mellitus as defined by fasting blood glucose >125 mg/dl or with ongoing treatment for Type 2 diabetes mellitus with the exception of insulin.

Exclusion Criteria:

* Women with a positive urine pregnancy test
* Body mass index >35 kg/m2
* Current daily long-acting insulin therapy (short acting, insulin as needed is not an exclusion).
* Clinical history of other major illness including cancer, renal failure, hepatic failure, or other conditions that in the judgment of the principal investigator make a clinical study inappropriate.
* Treatment with an investigational drug within the last twelve weeks
* History of a psychological illness or condition such as to interfere with the subject's ability to understand the requirements of the study.
* Treatment with vitamin E, vitamin C, and beta carotene, lipoic acid, and other food or herbal supplements within 1 month of enrollment. Subjects taking multivitamins or other forms of vitamin E and C in doses that do not exceed two times the recommended daily allowance will not be excluded.
* Recent change in diet or level of physical activity that in the judgment of the investigators would be likely to affect endothelial function (to be evaluated on a case by case basis).
* Ongoing illicit drug use or alcohol abuse.
* Sensitivity/intolerance to dietary polyols.

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2013-07-18 (Actual); Primary Completion 2014-12-01 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Endothelial function | 2 hours
  Change in pulse amplitude in the fingertip in response to reactive hyperemia measured by peripheral arterial tonometry.

CONTACTS AND LOCATIONS:
Overall Officials: Naomi M Hamburg, MD, Principal Investigator — Boston University
Locations (1):
- Boston University School of Medicine, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No